CLINICAL TRIAL: NCT01856881
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Multiple-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 876 in Subjects With Type 2 Diabetes
Brief Title: Multiple Ascending Dose Study in Subjects With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated on August 29th, 2014 due to a business decision by the Sponsor. The study was not terminated due to a safety reason.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20100018
Record Dates: First submitted 2013-03-25; First posted 2013-05-20 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 876 (Active Comparator)
  Interventions: Drug: AMG 876
- Placebo (Placebo Comparator)
  Interventions: Drug: AMG 876

INTERVENTIONS:
Drug: AMG 876 — Ascending multiple doses of study drug administered SC

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics following ascending multiple doses of AMG 876 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 to ≤ 65 years of age at the time of randomization
* Female subjects must be of documented non-reproductive potential
* Diagnosed with type 2 diabetes
* HbA1c ≥ 6.5% and ≤ 10%
* Fasting C-peptide value ≥ 0.8 ng/mL
* Body mass index (BMI) between ≥ 25.0 and ≤ 40.0 kg/m2 at screening

Exclusion Criteria:

* Female subjects who are lactating/breastfeeding or who plan to breastfeed while on study through 4 weeks after receiving the last dose of study drug.
* Male subjects with partners who are pregnant or planning to become pregnant while the subject is on study through 4 weeks after receiving the last dose of study drug
* Evidence or history at screening of diabetic complications with significant end-organ damage, eg, proliferative retinopathy and/or macular edema, estimated glomerular filtration rate < 60 mL/min/1.73m2 (calculated using the Modification of Diet in Renal Disease formula) or macroalbuminuria (ie, ≥ +1 proteinuria on urinalysis), diabetic neuropathy complicated by neuropathic ulcers, or severe autonomic neuropathy with gastroparesis, chronic diarrhea, or hypoglycemic unawareness
* Significant cardiac disease, including but not limited to, evidence or history of coronary artery disease, unstable angina, congestive heart failure, known arrhythmias of atrial or ventricular etiology, unexplained syncope, or syncope/seizures related to arrhythmia
* Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg) either on or off therapy at screening
* Triglycerides ≥ 500 mg/dL (5.64 mmol/L) at screening
* Hepatic liver enzymes ALT, AST, alkaline phosphatase (ALP), or total bilirubin (TBIL) levels > 1.5 times the upper limit of normal (ULN) at screening
* Fasting blood glucose > 270 mg/dL at the screening visit
* Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C virus antibodies (HepCAb)
* An unstable medical condition, defined as having been hospitalized within 28 days before day -1, major surgery within 6 months before day -1, or otherwise unstable in the judgment of the investigator (eg, risk of complications or adverse events unrelated to study participation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Subject incidence of treatment-emergent adverse events | 43 Days (Cohorts 1, 3, 5 and 7), 57 Days (Cohorts 2, 4, 6 and 9) or 71 Days (Cohort 8).
  Physical examinations, vitals, laboratory analytes, and ECGs
Subject incidence of anti-AMG 876 antibodies | 43 Days (Cohorts 1, 3, 5 and 7), 57 Days (Cohorts 2, 4, 6 and 9) or 71 Days (Cohort 8).
  Laboratory analytes

SECONDARY OUTCOMES:
AMG 876 serum PK parameters | 43 Days (Cohorts 1, 3, 5 and 7), 57 Days (Cohorts 2, 4, 6 and 9) or 71 Days (Cohort 8).
  Concentration-time profiles for AMG 876
Pharmacodynamic parameters | 43 Days (Cohorts 1, 3, 5 and 7), 57 Days (Cohorts 2, 4, 6 and 9) or 71 Days (Cohort 8).
  Concentration of fasting glucose, insulin, and C-peptide levels; Concentration-time profiles and AUC for metabolic parameters (eg, glucose, insulin, C peptide, glucagon, and non-esterified fatty acid concentrations); Fasting lipid levels (total cholesterol, low-density lipoprotein [LDL], high-density lipoprotein [HDL], and triglycerides); The following 7-point SMBG parameters: pre-meal average blood glucose, post-meal average blood glucose, 7-point average blood glucose, post-meal excursion, post-meal excursion average; Body weight, 24 hour weighted mean glucose(cohort 9 only)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (6):
  - Research Site, Chula Vista, California
  - Research Site, Miramar, Florida
  - Research Site, Overland Park, Kansas
  - Research Site, Cincinnati, Ohio
  - Research Site, San Antonio, Texas
  - Research Site, Renton, Washington

REFERENCES:
- [Derived] Kaufman A, Abuqayyas L, Denney WS, Tillman EJ, Rolph T. AKR-001, an Fc-FGF21 Analog, Showed Sustained Pharmacodynamic Effects on Insulin Sensitivity and Lipid Metabolism in Type 2 Diabetes Patients. Cell Rep Med. 2020 Jul 21;1(4):100057. doi: 10.1016/j.xcrm.2020.100057. eCollection 2020 Jul 21. PMID 33205064
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com